CLINICAL TRIAL: NCT07124546
Title: Development of Acceptance and Commitment Therapy for Cancer Distress Among Rural and Urban Patients With Hepatobiliary Cancers (ACT-HBC)
Brief Title: Acceptance and Commitment Therapy (ACT-HBC) for the Improvement of Cancer Distress in Patients With Hepatobiliary Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Carrie Bronars, PhD, LP, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-010916; NCI-2025-05221 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-010916 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Malignant Hepatobiliary Neoplasm
MeSH Terms: interventions — Acceptance and Commitment Therapy; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (ACT-HBC) (Experimental): Patients attend ACT-HBC telehealth group sessions over 2 hours QW for 8 weeks.
  Interventions: Behavioral: Acceptance and Commitment Therapy; Other: Questionnaire Administration; Other: Telemedicine

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Attend ACT-HBC telehealth group sessions
  Other Names: ACT
Other: Questionnaire Administration — Ancillary studies
Other: Telemedicine — Attend ACT-HBC telehealth group sessions
  Other Names: Telehealth

SUMMARY:
This clinical trial studies whether Acceptance and Commitment Therapy for patients with hepatobiliary cancers (ACT-HBC) can be used to help improve cancer distress. Patients with hepatobiliary cancer (HBC) often experience high levels of distress and reductions in quality of life. ACT-HBC is a behavioral intervention tailored to patients with HBC. It helps patients cope with difficult thoughts and emotions while staying connected to what matters most in life, which may be an effective way to improve cancer distress.

ELIGIBILITY:
Inclusion Criteria:

* HBC diagnosis
* Age >= 18 years
* Able to provide written informed consent
* Verbally endorse cancer distress
* Access to the internet
* Read and write in English
* Reside in the states of Iowa, Minnesota, or Wisconsin

Exclusion Criteria:

* Other psychological therapy that started =< 2 months prior to prospective enrollment
* Inability to actively participate in and learn from group therapy (e.g., active/uncontrolled psychotic symptoms, neurological condition, personality pathology) as determined by clinical judgement in Behavioral Medicine Program (BMP) consultation. Individual therapy or alternative group therapy will be offered to patients ineligible per this criterion
* HBC remission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | At 8 weeks
  The Institute for Healthcare Improvement 10-point Likert scale (0-10) asks: "Would you recommend this program to your friends and family?" A score ≥ 7 indicates high individual satisfaction. Program satisfaction is achieved if 50% of individuals meet this cut-off.
Patient session attendance (Feasibility) | At 8 weeks
  Feasibility will be determined by the number of patients attending ≥ 4 sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie A Bronars, PhD, LP, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials